CLINICAL TRIAL: NCT00755859
Title: Corticosteroids and Azathioprine Versus Corticosteroids Alone in IgA Nephropathy: a Randomized Controlled Trial.
Brief Title: "Steroids and Azathioprine Versus Steroids Alone in IgAN"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: A. Manzoni Hospital (Other)
Responsible Party: Claudio Pozzi, A. Manzoni Hospital, Lecco, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IgANSTAZA
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-08

CONDITIONS: IGA Nephropathy
Keywords: IgA nephropathy; steroids; azathioprine; chronic kidney disease progression; proteinuria
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria | interventions — Steroids; Azathioprine; Methylprednisolone Hemisuccinate; deltacortene; Adenosine Triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Six month steroid course plus azathioprine
  Interventions: Drug: steroids plus azathioprine
- 2 (Active Comparator): six month steroid course
  Interventions: Drug: steroids

INTERVENTIONS:
Drug: steroids plus azathioprine — methylprednisolone 1 g i.v. for three consecutive days at the beginning of months 1, 3 and 5, followed by oral prednisone 0.5 mg/kg every other day plus azathioprine 1.5 mg/kg/day for six months
  Other Names: solumedrol; deltacortene; azatioprina
  Arms: 1
Drug: steroids — methylprednisolone 1 g i.v. for three consecutive days at the beginning of months 1, 3 and 5, followed by oral prednisone 0.5 mg/kg every other day for six months
  Other Names: solumedrol; deltacortene
  Arms: 2

SUMMARY:
In a previous trial the investigators found that the effect of steroids in IgA nephropathy diminish over time. The difference in renal survival is striking up till the third year, but then remains constant. A six-month course of steroid therapy may be not enough to ensure a stable remission. The investigators hypothesized that a more aggressive treatment may obtain long-term better results. The investigators conducted a randomised controlled trial to assess the utility of low-dose azathioprine added to steroids in adult IgAN patients.

DETAILED DESCRIPTION:
In 1999, we published a multicenter, randomized, controlled trial, which compared a 6-month steroid course with supportive therapy in 86 patients with IgAN. After 5 years of follow-up, the risk of a 50% increase in plasma creatinine from baseline was significantly lower in the treated patients; proteinuria also decreased. However, the effect of steroids seemed to diminish over time. The difference in renal survival was particularly striking up till the third year, but then remained constant. We hypothesised that a six-month course of steroid therapy is not enough to ensure a stable remission, and a more aggressive treatment may be required to obtain long-term better results. At this regard, some studies of combined treatment with corticosteroids and azathioprine found that treatment was effective in preserving renal function and in reducing proteinuria. However, these studies did not clarify whether azathioprine added further benefit to steroids in the long term. We conducted a randomised controlled trial to assess the utility of low-dose azathioprine added to steroids in adult IgAN patients.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven IgA nephropathy
* creatinine ≤ 2.0 mg/dl for at least three months
* proteinuria ≥ 1.0 g/day for at least three months

Exclusion Criteria:

* treatment with steroids or cytotoxic drugs during the previous three years
* contraindications to steroids or azathioprine
* Henoch-Schöenlein purpura
* diabetes mellitus
* severe hypertension (diastolic blood pressure > 120 mmHg)
* lupus erythematosus systemicus
* malignancies
* active peptic-ulcer disease
* pregnancy
* viral hepatitis or other infections

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 1998-05; Primary Completion 2004-12 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
progression of renal disease, estimated by the time to 50% increase in plasma creatinine from baseline. | Every month for the first six months, then six months

SECONDARY OUTCOMES:
evolution of proteinuria over time | every months for the first six months and then every six months
safety | every months for the first six months and then every six months

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Pozzi, MD, Principal Investigator — A Manzoni Hospital, Lecco, Italy; Francesco Locatelli, MD, Study Chair — A Manzoni Hospital, Lecco, Italy; Simeone Andrulli, MD, Study Director — A Manzoni Hospital, Lecco, Italy; Antonello Pani, MD, Study Director — Hospital "G. Brotzu", Cagliari, Italy; Paolo Altieri, MD, Study Director — Hospital "G. Brotzu", Cagliari, Italy; Gian B Fogazzi, MD, Study Director — Hospital "Maggiore" IRCCS, Milan, Italy; Claudio Ponticelli, MD, Study Director — Hospital "Maggiore" IRCCS, Milan, Italy
Locations (28):
- Italy (27):
  - Hospital "Bolognini", Seriate, BG
  - Hospital "Spedali Civili", Brescia, Brescia
  - Hospital of Montichiari, Montichiari, Brescia
  - "G. Brotzu" Hospital, Cagliari, Cagliari
  - Hospital "Cannizzaro", Catania, Catania
  - Hospital "S.Anna", Como, CO
  - Hospital "Istituti Ospitalieri", Cremona, CR
  - Hospital "S.Marta e S.Venera",, Acireale, CT
  - Hospital "S.Vincenzo", Taormina, CT
  - Hospital "Careggi", Florence, Firenze
  - Hospital of University, Foggia, Foggia
  - Department of Nephrology and Dialysis, A. Manzoni Hospital, Lecco, LC
  - Hospital "Maggiore", Lodi, LO
  - Hospital "C. Poma", Mantova, Mantova
  - Hospital "Uboldo", Cernusco sul Naviglio, MI
  - Hospital of Desio, Desio, MI
  - Hospital "Maggiore" IRCCS, Milan, MI
  - Hospital "S. Francesco", Nuoro, Nuoro
  - Hospital "A.Segni", Ozieri, Nuoro
  - Hospital "V. Cervello", Palermo, Palermo
  - University Hospital, Parma, Parma
  - Fondazione Maugeri" IRCCS, Pavia, Pavia
  - CNR-IBIM, Reggio Calabria, Reggio Calabria
  - Hospital "S. Maria Nuova", Reggio Emilia, Reggio Emilia
  - Hospital of Sondrio, Sondrio, Sondrio
  - CMID, Torino, Torino
  - Hospital "Belcolle", Viterbo, Viterbo
- Inselspital, Bern, Switzerland

REFERENCES:
- [Background] Locatelli F, Pozzi C, Del Vecchio L, Andrulli S, Pani A, Fogazzi G, Altieri P, Ponticelli C. Combined treatment with steroids and azathioprine in IgA nephropathy: design of a prospective randomised multicentre trial. J Nephrol. 1999 Sep-Oct;12(5):308-11. PMID 10630693